CLINICAL TRIAL: NCT02925000
Title: A Phase I/IIa, Open Label, Dose-escalation Study Investigating the Safety, Tolerability, and Pharmacokinetics of Intravenous Liposomal Vinorelbine Tartrate Injection in Patients With Advanced Malignancy
Brief Title: Dose-escalation Study of Intravenous Liposomal Vinorelbine Tartrate Injection in Patients With Advanced Malignancy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Taiwan Liposome Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TLC178A1001
Record Dates: First submitted 2016-08-23; First posted 2016-10-05 (Estimated); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Cancer
Keywords: Advanced Malignancy; lymphoma; TLC178
MeSH Terms: conditions — Neoplasms; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TLC178 (Experimental): Liposomal Vinorelbine
  Interventions: Drug: TLC178

INTERVENTIONS:
Drug: TLC178 — TLC178
  Other Names: Liposomal Vinorelbine

SUMMARY:
This is a phase I/IIa, Open label, Dose-escalation Study Investigating the Safety, Tolerability, and Pharmacokinetics of Intravenous Liposomal Vinorelbine Tartrate Injection in Patients with Advanced Malignancy.

DETAILED DESCRIPTION:
Protocol No: TLC178A1001

Name of Finished Product: LipoVNB (Liposomal Vinorelbine Tartrate)

Title of Study:

Phase I/IIa, Open label, Dose-escalation Study Investigating the Safety, Tolerability, and Pharmacokinetics of Intravenous Liposomal Vinorelbine Tartrate Injection in Patients with Advanced Malignancy.

Study duration:

Every patient will have a treatment period of 4-week cycles until completion of 6 cycles, progression of disease or intolerance, withdrawal of consent or Investigator's judgment, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria

* Male or female, ≥18 years of age (≥20 years of age in Taiwan)
* Patients with histologically/cytologically confirmed solid tumor, or lymphoma including PTCL or CTCL.
* Malignancies for which there is no standard therapy, or previously treated locally advanced, refractory/relapsed or metastatic disease for which local curative surgery, curable radiotherapy, or satisfactory systemic anticancer therapy is no longer available
* Having at least one measurable tumor
* ECOG Performance Status of ≤2
* Women of childbearing potential must have a negative pregnancy test.

Exclusion Criteria

* Patient with untreated or inadequate controlled brain metastases.
* Prior systemic standard or investigational anticancer therapy, including target therapy, chemotherapy, immunotherapy within 28 days prior to the first dose of study drug. The above mentioned conditions which the Investigator considers there is no more drug effect, such as ≥5 half-lives are permitted
* Prior radiotherapy within 4 weeks before screening
* Prior autologous stem cell transplantation within 3 months of screening and allogeneic stem cell transplantation within 6 months of screening
* More than 5 lines of previous cytotoxic therapies. For patients of CTCL who failed romidepsin, more than 4 lines of previous therapies
* Major surgery within 4 weeks prior to first administration of study drug
* History of myocardial infarction, unstable angina or severe congestive heart failure (New York Heart Classification Class IV) or major stroke within 3 months prior to screening period
* Medical history of uncontrolled but clinically significant abnormal cardiac conduction abnormalities at electrocardiogram (ECG) at screening, any history or evidence of long QT syndrome or QTcF interval >450 msec for males and >470 msec for females (according to Fridericia's correction) at screening
* Known HIV infection; active hepatitis B or C without concurrent treatment
* Coexistence of any active and uncontrolled infection
* Poor vital organ function defined
* Uncontrolled and unstable concurrent medical condition including psychiatric disorders and alcohol/substance dependence/abuse that will jeopardize the safety of the patient, interfere with the objectives of the study, or affect the patient compliance with study requirements, as determined by the Investigator
* Known allergy or hypersensitivity to the study drug or its components
* Use of strong inhibitors or inducers of cytochrome P450 enzymes CYP3A4
* Pregnant or breast feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2020-10-06 (Actual); Study Completion 2020-10-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) determination | 4 weeks
  To determine the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) ofintravenous LipoVNB given every 4 weeks (Q4W) in patients with advanced malignancies.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) parameters of AUC (0-inf) calculated by plasma concentration of vinorelbine[ | from day 1 to day 29
  Area under the plasma concentration time curve from zero (predose) extrapolated to infinity
Pharmacokinetics (PK) parameters of AUC (0-inf) calculated by plasma concentration of majormetabolite, 4-O-deacetylvinorelbine | from day 1 to day 29
  Area under the plasma concentration time curve from zero (predose) extrapolated to infinity
Pharmacokinetics (PK) parameters of AUC(0 - last) calculated by plasma concentration ofvinorelbine | from day 1 to day 29
  Area under the plasma concentration time curve from zero (predose) to the time of the lastquantifiable concentration
Pharmacokinetics (PK) parameters of AUC(0 - last) calculated by plasma concentration of majormetabolite, 4-O-deacetylvinorelbine | from day 1 to day 29
  Area under the plasma concentration time curve from zero (predose) to the time of the lastquantifiable concentration
Pharmacokinetics (PK) parameters of Cmax calculated by plasma concentration of vinorelbine | from day 1 to day 29
  Maximum plasma concentration observed
Pharmacokinetics (PK) parameters of tmax calculated by plasma concentration of vinorelbine | from day 1 to day 29
  Time of Cmax
Pharmacokinetics (PK) parameters of tmax calculated by plasma concentration of major metabolite,4-O-deacetylvinorelbine | from day 1 to day 29
  Time of Cmax
Pharmacokinetics (PK) parameters of t1/2 calculated by plasma concentration of vinorelbine | from day 1 to day 29
  Apparent terminal half life
Pharmacokinetics (PK) parameters of t1/2 calculated by plasma concentration of 4-O-deacetylvinorelbine | from day 1 to day 29
  Apparent terminal half life
Pharmacokinetics (PK) parameters of MRT(0-inf) calculated by plasma concentration of vinorelbine | from day 1 to day 29
  Mean residence time extrapolated to infinity
Pharmacokinetics (PK) parameters of MRT(0-inf) calculated by plasma concentration of 4-O-deacetylvinorelbine | from day 1 to day 29
  Mean residence time extrapolated to infinity
Dose exposure relationship in patients with advanced malignancies treated with single and multipledoses of LipoVNB | up to 6 months
  single and multiple dose effect
Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | up to 6 months
  treatment related AE
Incidence of Treatment-Emergent Adverse Events | up to 6 months
  TEAE percentage
LipoVNB antitumor activity assessed by response rate | up to 6 months
  antitumor response rate
LipoVNB antitumor activity assessed by duration of response | up to 6 months
  antitumor efficacy
Progression free survival (PFS) of patients with advanced malignancies treated with LipoVNB | up to 6 months
  PFS

CONTACTS AND LOCATIONS:
Overall Officials: Carl Brown, Study Director — Taiwan Liposome Company
Locations (3):
- United States (2):
  - Karmanos Cancer Center, Detroit, Michigan
  - Montefiore Medical Center, The Bronx, New York
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No